CLINICAL TRIAL: NCT03784066
Title: Durvalumab (MEDI4736) Plus Tremelimumab in Resectable, Locally Advanced Squamous Cell Carcinoma of the Oral Cavity: a Window of Opportunity Study
Brief Title: Durvalumab With or Without Tremelimumab in Resectable Locally Advanced Squamous Cell Carcinoma of the Oral Cavity
Acronym: DUTRELASCO
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: AstraZeneca (Industry); European Organisation for Research and Treatment of Cancer - EORTC (Network); Vlaams Instituut voor Biotechnologie (VIB) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESR-16-12192; 2017-000577-36 (EudraCT Number)
Record Dates: First submitted 2018-10-31; First posted 2018-12-21 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Oral Cavity Squamous Cell Carcinoma
Keywords: squamous cell carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Squamous Cell | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Intervention Model Description: The primary objective is to evaluate the biological response in the tumor upon treatment with Durvalumab, and in parallel, with combination of Durvalumab and Tremelimumab.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- A (Active Comparator): Durvalumab
  Interventions: Drug: Durvalumab
- B (Active Comparator): Durvalumab + Tremelimumab
  Interventions: Combination Product: Durvalumab + Tremelimumab

INTERVENTIONS:
Drug: Durvalumab — All patients will be treated with postoperative radiotherapy (66 Gy in standard fractionation).
  In case of positive section margins or extracapsular extension, 3 cycles of cisplatin 100 mg/msq on days 1, 22, and 43 will be added to standard fractionation radiotherapy (66 Gy).
  Durvalumab monotherapy (1500 mg) will be administered via IV infusion day -14 and at the start of radiation therapy, with repeat administration every 4 weeks at fixed dose for a total of 6 cycles postoperative.
  Arms: A
Combination Product: Durvalumab + Tremelimumab — All patients will be treated with postoperative radiotherapy (66 Gy in standard fractionation).
  In case of positive section margins or extracapsular extension, 3 cycles of cisplatin 100 mg/msq on days 1, 22, and 43 will be added to standard fractionation radiotherapy (66 Gy).
  Durvalumab + Tremelimumab combination therapy: Tremelimumab (75 mg) will be administered via IV infusion day -14 and at the start of radiation therapy, with repeat administration every 4 weeks at fixed dose for a total of 3 cycles postoperative, Durvalumab (1500 mg) will be administered via IV infusion day -14 and at the start of radiation therapy, with repeat administration every 4 weeks at fixed dose for a total of 6 cycles postoperative.
  Arms: B

SUMMARY:
This is a randomized, open-label, prospective, pilot phase I/II study with focus on translational research and on the evaluation of the biological changes that are observed in sequential tumor tissue acquisition in patients with newly diagnosed advanced (stage IV) oral cavity SCC. Patients are treated with Durvalumab (arm A) or Durvalumab + Tremelimumab (arm B) after biopsy-confirmed diagnosis of locally advanced resectable SCCHN of the oral cavity. After surgery, the standard of care treatment is radiotherapy, and, depending on risk assessment concurrent cisplatin. Patients will be treated with Durvalumab (arm A) or Durvalumab and Tremelimumab (arm B) during six additional cycles, starting from day one of the postoperative radiotherapy.

DETAILED DESCRIPTION:
Durvalumab has shown activity in squamous cell carcinoma of the head and neck. Locally advanced resectable cancers of this type represent a challenge, as the majority of these patients still die from this disease in spite of surgery, radio- and chemotherapy.

Checkpoint inhibitors have recently proven to prolong life in recurrent/metastatic SCCHN, and several new molecules are currently tested in clinical trials in this indication, including PD-1, PD-L1, and CTLA-4 antibodies, either as single agent or in combination. These compounds might represent a valuable treatment for SCCHN patients in the adjuvant setting, given the favorable toxicity profile. Combination of Durvalumab (PD-L1 inhibition) and Tremelimumab (CTLA-4 inhibition) is currently tested in recurrent/metastatic head and neck cancer, and compared to Durvalumab as single agent, and to standard of care chemotherapy.

In this study both options, i.e. durvalumab as a single agent or Durvalumab in combination with Tremelimumab, will be tested in a randomized fashion. Randomization would be used to reduce selection bias, in a non-comparative study. Newly diagnosed patients with SCCHN of the oral cavity, will be treated with a single dose of Durvalumab with or without Tremelimumab two weeks before scheduled surgery.

When patients are first diagnosed with a resectable oral SCC, a biopsy is taken to confirm the diagnosis, and surgery is planned. This standard practice thus involves sequential tissue harvesting, both at the time of biopsy as well as the final resection specimen, making it possible to observe hallmarks of immune response when patients are treated once with Durvalumab with or without Tremelimumab after confirmation of the diagnosis on biopsy, but before surgery.

ELIGIBILITY:
Inclusion Criteria:

* Resectable locally advanced oral cavity SCC stage IV
* Newly diagnosed disease
* Age ≥18 years at the time of screening
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at enrollment
* No active second malignancy during the last five years except non melanomatous skin cancer or carcinoma in situ of the cervix
* No prior chemotherapy, radiotherapy or targeted therapy including PD-1, PD-L1 or CTLA-4 antibodies for SCCHN, including durvalumab or tremelimumab
* Availability of blood samples for Translational research
* Negative pregnancy test
* Normal organ function
* No participation in another interventional clinical trial in the preceding 30 days prior to randomization
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* Before patient registration, written informed consent must be given according to ICH/GCP, and national/local regulations
* Body weight > 30 kg

Exclusion Criteria:

* Histologically or cytologically confirmed head and neck cancer of any other primary anatomic location in the head and neck
* Receipt of other treatments for cancer within 30 days prior to first dose of study treatment
* Previous radiotherapy in the head and neck region
* Previous systemic therapy for SCCHN
* Current or prior use of immunosuppressive medication within 14 days before the first dose of their assigned IP.
* History of allogeneic organ transplantation
* Active or prior documented autoimmune or inflammatory
* Uncontrolled intercurrent illness
* Active relevant second malignancy during the last five years
* Mean QT interval corrected for heart rate ≥470 ms
* History of active primary immunodeficiency
* Active infection Receipt of live, attenuated vaccine within 30 days prior to the first dose of IP.
* Female patients of childbearing potential who are pregnant or breast-
* Known allergy or hypersensitivity to IP or any IP excipient
* Any condition that, in the opinion of the Investigator, would interfere with evaluation of the IP or interpretation of patient safety or study results
* Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP
* Metastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2025-03-24 (Estimated); Study Completion 2026-03-24 (Estimated)

PRIMARY OUTCOMES:
Evaluation of biological response in tumor tissue by means of difference in CD8 lymfocyte infiltration density | The first biopsy will be harvested as part of the diagnostic screening procedures between day 28 and 14 before surgery. The second biopsy will be harvest from the resection specimen on day 0. IP will be given exactly 14 days before surgery.
  Difference in CD8 infiltration density will be evaluated on Formalin-Fixed Paraffin-Embedded sections. Measurements will be done both visually by trained pathologists and quantitative on immunofluorescence panel.

SECONDARY OUTCOMES:
Imaging | After 14 days of treatment, prior to surgery
  RECIST v1.1 will be used to compare MRI images to preoperative imaging in order to non-invasively detect potential radiological changes induced by the investigated drug.
68Ga-CXCR-4 PET/MR (optional) | After 14 days of treatment, prior to surgery
  RECIST v1.1 will be used to compare MRI images (as part of the 68Ga-CXCR-4 PET/MR) to preoperative imaging in order to:
  * assess the correlation of metabolic 68Ga-CXCR-4 PET/MR with immune response in the tumor
  * identify an imaging technique able to detect immunologic activity that could serve as an imaging biomarker to select early those patients that may benefit from durvalumab with or without tremelimumab.
Locoregional control in days | Up to 2 years after surgery
  Patient follow up according to standard of care will include locoregional control, measured in days.
Time to treatment failure in days | Up to 2 years after surgery
  Patient follow up according to standard of care will include time to treatment failure, measured in days.
Overall survival in days | Up to 5 years after surgery
  Overall survival will be measured in days

CONTACTS AND LOCATIONS:
Overall Officials: Paul Clement, Prof., Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No